CLINICAL TRIAL: NCT04511975
Title: A Phase 1b Study Evaluating the Safety and Efficacy of IBI188 in Combination With Azacitidine in Subjects With Newly Diagnosed Higher Risk Myelodysplastic Syndrome (MDS)
Brief Title: A Study Evaluating the Safety and Efficacy of IBI188 in Combination With AZA in Subjects With Newly Diagnosed MDS
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: pause for further assessment and study adjustment
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI188A103
Record Dates: First submitted 2020-08-05; First posted 2020-08-13 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: MDS
Keywords: MDS
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IBI188 + azacitidine (Experimental): Participants will receive IBI188 in combination with azacitidine
  Interventions: Drug: IBI188; Drug: Azacitidine

INTERVENTIONS:
Drug: IBI188 — IBI188: 100 mg/mL, intravenous infusion once a week
Drug: Azacitidine — Azacitidine (VIDAZA) for Injection:100 mg per vial, subcutaneous injection will be administered for 7 days in each 28 day cycle
  Other Names: VIDAZA

SUMMARY:
This is an open-label, phase 1b study to evaluate the safety, tolerability and preliminary efficacy of IBI188 in combination with Azacitidine in newly diagnosed higher risk MDS patients.

ELIGIBILITY:
Main Inclusion Criteria:

1. Newly diagnosed MDS subjects with higher risk.
2. Age ≥ 18 years old.
3. Eastern Cooperative Oncology Group score of 0-2.
4. Adequate organ function.
5. Subjects should take effective contraceptive measures.
6. Must sign the Informed Consent Form (ICF), and be able to follow all study procedures.

Main Exclusion Criteria:

1. Subject who has transformed from MDS to AML.
2. MDS subjects with lower risk.
3. Subjects who have received chemotherapy.
4. History of chronic hemolytic anemia
5. Prior exposure to any anti-CD47 or anti-SIRPα agents.
6. Subjects participating in another interventional clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-04-04 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 28 days
  Adverse events according to national Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 or customized AE severity grading as defined in the protocol
Efficacy of IBI188 in combination with AZA | 28 days
  International Working Group (IWG) 2006 criteria will be used to evaluate efficacy of IBI188 in combination with AZA for response criteria for MDS

CONTACTS AND LOCATIONS:
Overall Officials: Yi Luo, Study Director — Innovent Biologics
Locations (3):
- United States (3):
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - New Jersey Center for Cancer Research, Brick, New Jersey
  - Gabrail Cancer Center, Canton, Ohio